CLINICAL TRIAL: NCT01627236
Title: Efficacy of Short-term Immunosuppressive Therapy and Anti-allergenic Therapy in Severe Acute Exacerbation of Chronic Hepatitis B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe-bin Wu, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: zssywzb01
Record Dates: First submitted 2012-06-10; First posted 2012-06-25 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-08

CONDITIONS: Severe Acute Exacerbation of Chronic Hepatitis B
MeSH Terms: interventions — Methylprednisolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- glucocorticoid treatment group (Experimental)
  Interventions: Drug: methylprednisolone
- conventional treatment (No Intervention)

INTERVENTIONS:
Drug: methylprednisolone — methylprednisolone 1mg/kg intravenous drip qd，for 3 days glucocorticoid
  Arms: glucocorticoid treatment group

SUMMARY:
The investigators will investigate the clinicopathological features of chronic hepatitis B patients with severe exacerbation selected by uniform criteria, and treated with early introduction or reintroduction of corticosteroids and anti-allergenic therapy, in order to clarify the benefits and limitations of the effects of corticosteroids and anti-allergenic therapy for amelioration of clinically severe exacerbation of chronic hepatitis B. The investigators also observe the immune index in the change before and after the treatment, in order to searching for some prognostic index.

ELIGIBILITY:
Inclusion Criteria:

* serum hepatitis B surface antigen(HBsAg) positive for at least 6 months;
* All patients had a poor general condition, manifested as general malaise, fatigue, jaundice and so on;
* serum T-Bil of 85.5 mmol/L or more; or serum T-Bil rises 17.1 mmol/L or more per day; or PTA of less than 60%;
* serum ALT of 20 times or more the ULN.

Exclusion Criteria:

* superinfection or co-infection with hepatitis A, C, D, E, cytomegalovirus and HIV, or Epstein-Barr virus;
* other liver diseases such as alcoholic liver disease, drug-induced hepatitis, Wilson disease and autoimmune hepatitis;
* ascites or gastrointestinal bleeding or peptic ulcer or esophageal varix by electronic gastroscope examination;
* decompensated liver cirrhosis;
* severe bacterial or fungal infections;
* a history of diabetes or cardiac disease or hypertension or nephrosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-08 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
survival rate | eight weeks
liver function | eight weeks
  ALT,albumin,bilirubine,
HBV-DNA | eight weeks
prothrombin activity | eight weeks
Child-Pugh degree | eight weeks
model for end-stage liver disease | eight weeks

SECONDARY OUTCOMES:
length of patient stay | eight weeks
hospitalization costs | eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-liang Gao, professor, Study Director — Deparment of Infectious Diseases, the Third Affiliated Hospital of Sun Yat-sen University
Locations (1):
- Deparment of Infectious Diseases, the Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China